CLINICAL TRIAL: NCT03466814
Title: ORENCIA Safety Surveillance in Japanese Children and Adolescents With Active Juvenile Idiopathic Arthritis (JIA)
Brief Title: Study of the Safety of Orencia in Japanese Children and Adolescents With Active Juvenile Arthritis of Unknown Origin
Status: Completed | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: IM101-635
Record Dates: First submitted 2018-03-09; First posted 2018-03-15 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Undifferentiated Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- JIA participants
  Interventions: Other: Non-Interventional

INTERVENTIONS:
Other: Non-Interventional — Non-Interventional

SUMMARY:
Observational study of abatacept in the treatment of JIA in Japan.

ELIGIBILITY:
Inclusion Criteria:

* All JIA participants who initiate treatment with Orencia in accordance with the prescribing information

Exclusion Criteria:

* Participants receiving Orencia for an off-label indication

Other protocol defined inclusion/exclusion criteria could apply

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study is a local, prospective, non-interventional, non-controlled, multicenter, observational study for authorization of abatacept in the treatment of JIA
Sampling Method: Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2018-04-06 (Actual); Primary Completion 2021-07-21 (Actual); Study Completion 2021-07-21 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | 1 year

SECONDARY OUTCOMES:
Safety measured by number of participants who receive at least 1 dose of Orencia | 1 year
Efficacy measured by number of participants who receive at least 1 dose of Orencia | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Shinjuku-ku, Tokyo, Japan

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm